CLINICAL TRIAL: NCT05009121
Title: The Reliability of the Box and Block Test in People After Stroke
Status: Active, not recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Rybářová, occupational therapist, Charles University, Czech Republic
Other Study IDs: 75/21 S-IV
Record Dates: First submitted 2021-08-12; First posted 2021-08-17 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Motor Activity
Keywords: standardized test; occupational therapy; fine motor skills; Box and Block Test; inter-rater reliability; variability; Czech language; Stroke
MeSH Terms: conditions — Motor Activity; Stroke | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Czech adult people after stroke: Czech adult people after stroke will be asked basic questions about present feelings according to their condition using a questionnaire. Then they will be tested by the Box and Block Test in only one session. Video of their performance will be obtained. The Box and Block Test will be done during their regular rehabilitation by occupational therapist.
  Interventions: Diagnostic Test: Box and Block Test

INTERVENTIONS:
Diagnostic Test: Box and Block Test — At first, each person will be asked basic questions about present feelings according to their condition using a questionnaire. Than he/she will be tested by the Box and Block Test according to the Czech version of extended manual for this test in only one session. Audio recording of verbal instructions will be used.
  The results will be used only for establishing of the variability and inter-rater reliability of the Box and Block Test, not for patients' other interventions.
  Other Names: questionnaire

SUMMARY:
The main aim of the pilot project is to establish inter-rater reliability, internal variability and variability of results got in Box and Block Test administered according to the new Czech extended version of its manual.

DETAILED DESCRIPTION:
New Czech manual for the Box and Block Test was made by back-translation method. It was updated and extended by new rules for unification of it´s performing. The manual include instructions for performing three trials.

At least 20 adult people after stroke will be tested by this test according to this new Czech manual. Video of patients' performance will be obtained.

The inter-rater reliability, internal variability and variability of results will be established.

ELIGIBILITY:
Inclusion Criteria:

* Czech language as a mother tongue
* Adult (age 18 and more)
* Patient after Stroke attending the Department of Rehabilitation Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague
* Able to move 25mm X 25mm block at least by 10 cm
* Able to complete testing with full 3 attempts
* Able to sit for 20 minutes

Exclusion Criteria:

* use of drugs affecting attention
* vision impairment uncorrectable with glasses
* severe hearing loss
* inability to understand instructions
* inability to complete testing
* failure to sign Informed consent for probation with inclusion to research and Consent to the collection and processing of personal data during the study at the General University Hospital in Prague

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — based on self-representation
Study Population: Czech adult people after stroke
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
results from the Box and Block Test | 30 minutes
  number of transported blocks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, First Faculty of Medicine, Charles University and General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No